CLINICAL TRIAL: NCT00619840
Title: Placebo-Controlled Multi-Centre Double-Blind Trial for Adults With Extended-Release Methylphenidate for ADHD
Acronym: EMMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medice Arzneimittel Pütter GmbH & Co KG (Industry)
Responsible Party: Dr. Roland Fischer/Head of Medical Dept., Medice Arzneimittel Pütter GmbH & Co. KG
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6520-9979-06
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2008-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Attention Deficit Hyperactivity Disorder; adult; methylphenidate hydrochloride; Medikinet retard; long-term observation; controlled clinical trial; safety; randomized, double-blind, placebo-controlled trial; treatment; central nervous system stimulants; therapeutic uses
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: methylphenidate hydrochloride
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: methylphenidate hydrochloride — sustained release, 10 mg capsule 1-3 capsules twice daily according to an individual titration schedule
  Other Names: Medikinet retard
  Arms: 1
Drug: Placebo — 10 mg capsule 1-3 capsules twice daily according to an individual titration schedule
  Arms: 2

SUMMARY:
Investigation of efficacy and tolerability of extended-release MPD in adults with ADHD, compared with a placebo, and to acquire knowledge through long-term observation of adults

ELIGIBILITY:
Inclusion Criteria:

* Patient treated as outpatient or inpatient
* Patient has a good command of German
* Score of 85 or greater in the IQ test (MWT-B)
* Diagnosis of ADHD according to ADHD-CL (DSM IV) and WRI-WRAADDS > 28 points
* ADHD symptoms have existed since childhood (WURS-k >= 30)
* Body mass index >= 20
* Willing to eat breakfast
* Patient is willing and able to come to the observation appointments
* Written consent of the patient to participate in the study

Exclusion Criteria:

* Treatment with psychostimulants in the past 2 weeks
* Inconsistencies in the CAARS- S:L >= 8 (Inconsistency Index)
* Shift work or night work
* Alcohol, medication or drug dependency in the past 6 months or manifest drug abuse
* Diagnosis of a psychosis (SKID-I)
* Epileptic attacks in the past
* EEG results which suggest epilepsy
* Clinically relevant liver disease
* Clinically relevant hyperthyroidism (relevantly elevated TSH, T4)
* Acute depressive episode according to ICD-10 F32.2 and ICD-10 32.3 (SKID-I)
* Illnesses with schizophrenic symptoms (SKID-I)
* Acute manic episode, bipolar disorder (SKID-I)
* Diagnosis of a tic disorder
* Acute anorexia
* Acute prominent panic disorder and generalised anxiety (SKID-I)
* Clinically relevant kidney disorders
* Known high blood pressure
* Known occlusive arterial disease
* Known angina pectoris
* Known coronary heart disease and state after myocardial infarction
* Known tachycardial arrhythmias
* Post-stroke status
* Known elevated intra-occular pressure
* Known enlarged prostates
* Participation in a clinical study within the past 30 days
* Participation in this study at an earlier point in time
* Simultaneous participation in another clinical trial
* Women of child-bearing age without adequate contraception
* Patients with terminal illness (e.g. cancer)
* Pregnancy (positive pregnancy test) or lactation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2004-11; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
German validated version of the WRAADDS: Wender-Reimherr-Interview (WRI) | Week 24

SECONDARY OUTCOMES:
CAARS self report: long version (CAARS-S:L) | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rösler, Prof. Dr., Principal Investigator — Institute of Forensic Psychology and Psychiatry, University of Saarland
Locations (1):
- Institute of Forensic Psychology and Psychiatry, Homburg/Saar, Saarland, Germany